CLINICAL TRIAL: NCT00119340
Title: Fludarabine and Low-Dose TBI Dose Escalation to Determine the Optimal Regimen for Achieving High Rates Engraftment of Unrelated Donor Peripheral Blood Stem Cell in Patients With Chronic Myeloid Leukemia - A Multi-Center Trial
Brief Title: Fludarabine, Total-Body Irradiation, and Donor Stem Cell Transplant Followed By Cyclosporine and Mycophenolate Mofetil in Treating Patients With Chronic Myelogenous Leukemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Brenda Sandmaier, Fred Hutchinson Cancer Research Center
Purpose: Treatment
Other Study IDs: 1939.00; FHCRC-1939.00; CDR0000432959 (Registry Identifier: PDQ)
Record Dates: First submitted 2005-07-12; First posted 2005-07-13 (Estimated); Last update posted 2010-09-21 (Estimated); Status verified 2010-09

CONDITIONS: Leukemia
Keywords: accelerated phase chronic myelogenous leukemia; Philadelphia chromosome positive chronic myelogenous leukemia; relapsing chronic myelogenous leukemia; chronic phase chronic myelogenous leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Accelerated Phase; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Myeloid, Chronic-Phase | interventions — Cyclosporine; fludarabine phosphate; Mycophenolic Acid; Peripheral Blood Stem Cell Transplantation; Radiotherapy

INTERVENTIONS:
Drug: cyclosporine
Drug: fludarabine phosphate
Drug: mycophenolate mofetil
Procedure: peripheral blood stem cell transplantation
Radiation: radiation therapy

SUMMARY:
RATIONALE: Giving low doses of chemotherapy, such as fludarabine, and radiation therapy before a donor stem cell transplant helps stop the growth of cancer cells. It also stops the patient's immune system from rejecting the donor's stem cells. The donated stem cells may replace the patient's immune system and help destroy any remaining cancer cells (graft-versus-tumor effect). Sometimes the transplanted cells from a donor can also make an immune response against the body's normal cells. Giving cyclosporine and mycophenolate mofetil after transplant may stop this from happening.

PURPOSE: This phase I/II trial is studying the side effects and best dose of fludarabine, total-body irradiation, and donor stem cell transplant followed by cyclosporine and mycophenolate mofetil and to see how well they work in treating patients with chronic myelogenous leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine whether increasing the intensity of a nonmyeloablative conditioning regimen comprising fludarabine and total body irradiation allows achievement of a donor T-cell chimerism level of > 40% on day 28 post-transplantation in 90% or more of patients with chronic myelogenous leukemia undergoing allogeneic peripheral blood stem cell transplantation and immunosuppression comprising cyclosporine and mycophenolate mofetil.
* Determine the feasibility of reducing the day 84 graft rejection rate/graft failure to < 10% in patients treated with this regimen.
* Determine the feasibility of maintaining the incidence of grade 4 acute graft-versus-host disease at < 10% in patients treated with this regimen.
* Determine the feasibility of maintaining the day 200 nonrelapse mortality rate at < 15% in patients treated with this regimen.

Secondary

* Determine the rate of complete cytogenetic remission in patients treated with this regimen.
* Determine the probability of actuarial disease-free survival of patients treated with this regimen.
* Determine the pharmacokinetics of mycophenolate mofetil and fludarabine in these patients.

OUTLINE: This is a multicenter, dose-escalation study of fludarabine and total-body irradiation (TBI).

* Nonmyeloablative conditioning regimen: Patients receive fludarabine IV on days -4 to -2 OR days -6 to -2. Patients undergo TBI on day 0.
* Allogeneic peripheral blood stem cell transplantation (PBSCT): After the completion of TBI, patients undergo allogeneic PBSCT on day 0.
* Immunosuppression: Patients receive oral cyclosporine twice daily on days -3 to 100 followed by a taper to day 177 in the absence of graft-versus-host disease (GVHD). Beginning within 4-6 hours after the completion of PBSCT, patients receive oral mycophenolate mofetil 2-3 times daily on days 0-40 followed by a taper to day 96 in the absence of GVHD.

Cohorts of 5-25 patients receive cumulative doses of fludarabine and escalating doses of TBI until 2 of 5, 3 of 10-15, 4 of 20, or 5 of 25 patients experience a day 28 post-transplant T-cell chimerism level ≤ 40% and/or a day 84 post-transplant graft rejection rate of > 10%.

After completion of study transplantation, patients are followed 3 times weekly for 3 months, at 6, 12, and 18 months, annually for 5 years, and then periodically thereafter.

PROJECTED ACCRUAL: A total of 5-75 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of chronic myelogenous leukemia (CML), meeting 1 of the following criteria:

  * First or second chronic phase

    * Philadelphia chromosome-positive (Ph+) disease by cytogenetics or fluorescent in situ hybridization (FISH)
  * First accelerated phase, meeting any of the following criteria:

    * More than 10% but < 30% myeloblasts and promyelocytes in bone marrow or peripheral blood
    * Any additional clonal cytogenetic abnormalities
    * Increasing splenomegally
    * Extramedullary tumor
    * WBC, platelet count, or hematocrit pertubations not controlled by therapy with hydroxyurea, interferon, or imatininb mesylate
    * Persistent unexplained fever or bone pain
* Less than 5% blasts in marrow at time of transplant

  * No blast crisis
* No other curative therapy exists
* Received prior imatinib mesylate AND meets ≥ 1 of the following criteria:

  * Hematologic evidence of disease progression
  * Lack of complete hematologic response after 3 months of treatment with imatinib mesylate
  * Cytogenetic evidence of disease progression, defined as an increase in Ph+ cells or BCR/ABL-positive (BCR/ABL+) cells of > 25%
  * Lack of complete cytogenetic remission (no Ph+ cells by cytogenetic analysis or BCR/ABL+ cells by FISH) after 1 year of treatment with imatinib mesylate
  * At least 65% Ph+ cells by cytogenetic analysis or BCR/ABL+ cells by FISH after 6 months of treatment with imatinib mesylate
  * Less than 3-log reduction in BCR/ABL mRNA levels by quantitative polymerase chain reaction (Q-PCR) compared to a standard baseline level after 1 year of treatment with imatinib mesylate
  * Molecular evidence of disease progression, defined as > 1 log increase in BCR/ABL mRNA levels by Q-PCR, detected in 2 samples
  * Experienced adverse events with imatinib mesylate treatment that would preclude further administration of the drug
  * Patient refused further treatment with imatinib mesylate despite lack of disease progression
* Refused conventional myeloablative allogeneic stem cell transplantation OR at high risk for regimen-related toxicity due to pre-existing medical conditions (for patients < 50 years of age)
* Unrelated donor available

  * Matched at HLA-A, -B, -C, -DRB1, and -DQB1 by high-resolution typing

    * A single allele* disparity for HLA-A, -B, or -C allowed
  * Negative anti-donor cytotoxic crossmatch
  * Not a marrow donor NOTE: *Patient and donor pairs homozygous at a mismatched allele (e.g., the patient is A*0101 and the donor is A*0201) are considered a two-allele mismatch and are not allowed
* No CNS involvement with disease that is refractory to intrathecal chemotherapy

PATIENT CHARACTERISTICS:

Age

* Any age

Performance status

* Karnofsky 70-100%
* Lanksy 50-100% (for pediatric patients)

Life expectancy

* Not specified

Hematopoietic

* See Disease Characteristics

Hepatic

* No fulminant liver failure
* No cirrhosis of the liver with evidence of portal hypertension
* No alcoholic hepatitis
* No esophageal varices
* No history of bleeding esophageal varices
* No hepatic encephalopathy
* No uncorrectable hepatic synthetic dysfunction evidenced by prolongation of PT
* No ascites related to portal hypertension
* No bacterial or fungal liver abscess
* No biliary obstruction
* No chronic viral hepatitis AND bilirubin > 3 mg/dL
* No symptomatic biliary disease

Renal

* Not specified

Cardiovascular

* Ejection fraction ≥ 40%
* No cardiac failure requiring therapy
* No poorly controlled hypertension (i.e., blood pressure ≥ 150/90 mm Hg despite standard medication)

Pulmonary

* DLCO ≥ 35% (corrected)
* No requirement for supplementary continuous oxygen
* Pulmonary nodules allowed at the discretion of the principal investigator

Immunologic

* HIV negative
* No uncontrolled systemic infection
* No fungal infection with radiological progression after treatment with amphotericin B or active triazole for > 1 month

Other

* Not pregnant or nursing
* Fertile patients must use effective contraception during and for 12 months after completion of study treatment
* No other active malignancy except nonmelanoma skin cancer
* No prior localized malignancy at high risk (≥ 20%) of recurrence

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics
* See Chemotherapy

Chemotherapy

* See Disease Characteristics
* More than 3 weeks since prior cytotoxic chemotherapy

  * Imatinib mesylate and interferon are not considered cytotoxic chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2005-04; Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Increase number of patients with donor T-cell chimerism from > 40% to 90% on day 28 post-transplant
Reduce graft rejection rate to < 10% day 84 post-transplant
Maintain acute graft-vs-host disease (GVHD) incidence of 10%
Maintain nonrelapse mortality incidence of < 15% on day 200 post-transplant

SECONDARY OUTCOMES:
Rate of complete cytogenetic remission
Probability of actuarial disease-free survival
Pharmacokinetics

CONTACTS AND LOCATIONS:
Overall Officials: Brenda Sandmaier, MD, Principal Investigator — Fred Hutchinson Cancer Center
Locations (3):
- United States (3):
  - Veterans Affairs Medical Center - Seattle, Seattle, Washington
  - Seattle Cancer Care Alliance, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington